CLINICAL TRIAL: NCT03569943
Title: Implantation of Trans-tympanic Aerator Using a Robotic Microsurgical Assistance Tool
Brief Title: Robot Based Tympanic Tube Placement
Acronym: ROBOTOL
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in medical practice on the management of the eligible population
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: P160408J; 2017-A03159-44 (Other: ANSM)
Record Dates: First submitted 2018-06-15; First posted 2018-06-26 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Patient Operated on From a Vestibular Schwannoma With a Middle Ear Exclusion
Keywords: Robot based procedure; RobOtol; Tympanic drain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Robotol (Experimental)
  Interventions: Device: Robot Based Transtympanic drain placement

INTERVENTIONS:
Device: Robot Based Transtympanic drain placement — Placement of a transtympanic drain with a robot based device assistance called RobOtol

SUMMARY:
Middle ear surgery is performed in a deep workspace through a narrow approach to the tympanic cavity, either by the external auditory canal, or by drilling the temporal bone. It uses thin and long instruments as a delicate and precise gesture on the ossicular chain or manipulation of very light prostheses is necessary. The results of middle ear procedures relies upon the surgeon experience and his gesture accuracy. For this reason, a robot-based device designed to assist the surgeon during middle ear procedure has been build. The goal of the present protocol is to evaluate the robot in a simple procedure to ensure its safety before using the device in more complex cases.

The precision of the robot during transtympanic tube placement will be evaluated. The following benefits are expected:

* Significantly reduced risk of transtympanic tube on the other side of the eardrum.
* Positioning of the transtympanic tube in the desired tympanic quadrant
* Reduces the size of the entry point to prevent tearing
* Reduced risk of injury to the external auditory canal

Once the safety of use of the robot is demonstrated in this protocol, the goal will be to evaluate it later in more complex surgical gestures in other protocols. The future application of the robot will be the placement of middle ear implant prosthesis in the context of the surgery for cholesteatoma, otosclerosis or insertion of cochlear implants.

DETAILED DESCRIPTION:
Description of the population to be studied and justification of its choice:

This study is going to include a single group of patients presenting a vestibular schwannoma that will benefit from an removal by translabyrinthine approach with exclusion from the middle ear under general anesthesia. During this surgery, the tympanic membrane is systematically sacrificed and the inner ear opened with as consequence a complete loss of residual hearing and vertigo for a few days. In this protocol research, the patients will participate by accepting an robot based placement of a tympanic ventilation drain during the surgery before the sacrifice of the tympanic membrane.

All the patients will be adults, living in France, benefiting from the cover of the French health care system. The people participating to the research will have to give their consent to participate to the study.

Name and brief description of one or several experimental medical devices:

The concept of the device RobOtol® is based on a teleoperated system with 6 degrees of freedom.

The medical device is European Conformity (CE) marked since in June, 2016. The team of Ear, Nose and Throat (ENT) of Pitié-Salpêtrière (PSL) university hospital will lead this project.

Description and justification of the methods and the duration of study:

The studied device is a drain mounted on a trocar placed by means of the teleoperated system RobOtol.

The gold standard device and procedure is a drain inserted by the surgeon with forceps after incision of the eardrum.

The equipment RobOtol will be driven by the surgeon. The procedure will be conducted under general anesthesia.

Summarize of predictable and known benefits and risks for the people participating to the study:

There is no individual expected benefit considering the choice of the included population in the protocol. The population was chosen to eliminate the risks of unwanted effect during the installation of the drain by the robot (in particular the risks for the tympanic membrane).

The patients presenting an indication of tympanic ventilation drain placement (ex: serous otitis), have the exceptional risks, a hearing loss, a secondary infection of the drain or vertigo, or facial palsy.

The population chosen in this study has to benefit from a removal of a vestibular schwannoma. Within the procedure of this surgery, a total loss of the hearing, a sacrifice of the tympanic membrane and vertigo are expected and predictable consequences of the surgical technique. For that reason, there is no additional risk of complication.

The only risk is the fact that the general anesthesia will be prolonged for the study, for approximately 15 min on a surgery requiring an average duration of anesthesia of 5,5 hours (1 hour of perioperative anesthesia, 4,5 hours of surgery).

PROGRESS OF THE SEARCH

Modalities(Methods) of recruitment:

Fifteen adults presenting a vestibular schwannoma that will benefit from a removal by translabyrinthine approach with exclusion from the middle ear under general anesthesia will be included after information and obtaining of their written consent.

1. Visit of selection and inclusion The recruitment of the patients will be made from the line of the new patients by the investigators for the consultation of ENT of PSL.

   Visit of selection / inclusion in the study by the ENT ( D0):

   O Clinical examination: otoscopy, check of the diameter of the external auditory canal o Check of the criteria of inclusion and non inclusion o Information of the patient o Signature of the informed consent by the patient o Collection clinical data: sex, age, operated side (left / right), previous otological history, diameter of the external auditory canal
2. Visit of follow-up of the study

   The intervention by the ENT (D14):

   The intervention will take place in the operating room of the building Babinski and the service of ENT;
3. Visit of the end of the research There is no visit of post-operative follow-up nor visit of the end of planned research.

The patient sees his participation in the research ending after the removal of the tympanic membrane at D0.

ELIGIBILITY:
Inclusion Criteria:

* Patient candidate for exclusion of the middle ear when performing a translabyrinthine approach during a vestibular schwannoma surgery
* Patient over 18 years old

Exclusion Criteria:

* Patient with psychomotor retardation or behavioral problems that preclude clinical examination
* Patient with an external auditory canal diameter of less than 3 mm
* Patient participating in another interventional clinical trial
* Breastfeeding or pregnant woman
* Patient not residing in France
* Patient under tutorship / guardianship or under security measure
* Patient who has not signed a written consent
* Patient not benefiting from french national health insurance system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Drain position on the tympanic membrane | one day
  Video recording of the procedure and tympanic membrane collection and microscopic analysis will used to assess drain position

SECONDARY OUTCOMES:
The occurence of a bleeding intraoperative from the eardrum or from the external auditory canal | one day
  Video recording of the procedure will used to assess this measure Yes/no answer
The occurence of a lesion of the tympanic membrane except the section necessary for the placement of the drain (tympanic perforation, accidental tear) | one day
  Video recording of the procedure and tympanic membrane collection and microscopic analysis will used to tympanic lesions
The number of contact between the cutaneous cover of the external auditory canal and the instrument of the robot | one day
  Video recording of the procedure will used to assess this measure (number of contacts)
Duration of installation of the robot and the procedure | one day
  Duration of installation of the robot and the procedure will be collected

IPD SHARING:
Plan to Share IPD: No